CLINICAL TRIAL: NCT07189975
Title: Effects and Comparison of Eccentric Cycling Trainings Versus Concentric Cycling Training on Muscular and Functional Capacities in Sedentary People
Brief Title: Eccentric Cycling : a Promising Training Modality for Sedentary People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Vandenbroeck Benoit, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B7072023000019 - 2023/72
Record Dates: First submitted 2025-08-25; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Sedentary; Deconditioning; Eccentric Exercise Training; Eccentric Cycling Exercise; Elderly; Healthy Participants
Keywords: Eccentric cycling; Sedentarity; Elderly; Physical deconditioning; Training modality; Rehabilitation; Eccentric training
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric Interval (Experimental): Participants in this arm had to follow a high intensity interval training using an eccentric ergocycle
  Interventions: Other: High intensity eccentric cycling training
- Eccentric continuous (Experimental): Participants in this arm had to follow a moderate intensity continuous training using an eccentric ergocycle
  Interventions: Other: Moderate intensity eccentric cycling training
- Concentric interval (Experimental): Participants in this arm had to follow a high intensity interval training using a concentric ergocycle
  Interventions: Other: High intensity concentric cycling training

INTERVENTIONS:
Other: High intensity eccentric cycling training — This intervention is a high intensity interval training using an eccentric ergocycle
  Arms: Eccentric Interval
Other: Moderate intensity eccentric cycling training — This intervention is a moderate intensity continuous training using an eccentric ergocycle
  Arms: Eccentric continuous
Other: High intensity concentric cycling training — This intervention is a high intensity interval training using a concentric ergocycle
  Arms: Concentric interval

SUMMARY:
The present study aims to compare the acute and training responses of (1) eccentric high intensity interval training (EI), (2)work-matched continuous eccentric training (EC), and (3) concentric high intensity interval training (CI), all performed on cycle ergometers. The variables of interest include ratings of perceived exertion (RPE), cognitive demand (Fat), heart rate (HR), maximal oxygen consumption (VO₂max), maximal aerobic power (MAP), and various functional and health-related parameters.

It is hypothesized that eccentric interval training will produce comparable or superior improvements in functional outcomes relative to concentric interval training, but at a lower metabolic and perceptual cost. Furthermore, eccentric interval training is expected to yield greater physiological benefits than continuous eccentric training for a similar perceived and metabolic load.

Forty-three sedentary healthy adults (23 men and 20 women) were recruited for this study based on predefined inclusion and exclusion criteria. Participants were randomly (stratified randomization) allocated into one of three training groups.

Participants attended the laboratory on 28 occasions over a 14-week period, with two sessions per week.

Participants in the EI and EC groups trained using an eccentric ergometer, while the CI group trained on a concentric ergometer. Baseline and post-intervention assessments were conducted during weeks 1 and 14, respectively. These included a maximal incremental cycling test to determine VO₂ peak and concentric MAP, followed by six functional performance assessments.

DETAILED DESCRIPTION:
The present study aims to compare the acute and training responses of (1) eccentric HIIT, (2)work-matched continuous eccentric training, and (3) concentric HIIT, all performed on cycle ergometers. The variables of interest include ratings of perceived exertion (RPE), cognitive demand (Fat), heart rate (HR), maximal oxygen consumption (VO₂max), maximal aerobic power (MAP), and various functional and health-related parameters.

It is hypothesized that eccentric HIIT will produce comparable or superior improvements in functional outcomes relative to concentric HIIT, but at a lower metabolic and perceptual cost. Furthermore, eccentric HIIT is expected to yield greater physiological benefits than continuous eccentric training for a similar perceived and metabolic load.

Forty-three healthy adults (23 men and 20 women) were recruited for this study based on predefined inclusion and exclusion criteria. Participants were randomly (stratified randomization) allocated into one of three training groups:

* Eccentric Interval Group (EI): n = 15 (8 men, 7 women); age = 62.6 ± 3.9 years old (yo)
* Eccentric Continuous Group (EC): n = 15 (8 men, 7 women); age = 61.6 ± 6.3 yo
* Concentric Interval Group (CI): n = 13 (7 men, 6 women); age = 60.5 ± 5.1 yo All participants were unaccustomed to eccentric cycling and engaged in no more than 2 hours of recreational physical activity per week. Individuals with recent lower limb injuries or chronic medical conditions were excluded. Prior to participation, all individuals were fully informed of the study procedures, potential risks, and provided written informed consent. The study protocol received ethical approval from the Ethics Committee of the University of Liège (Ref. 2023/72), and all procedures conformed to the Declaration of Helsinki.

Participants in the EI and EC groups trained using an eccentric ergometer, while the CI group trained on a concentric ergometer. Baseline and post-intervention assessments were conducted during weeks 1 and 14, respectively. These included a maximal incremental cycling test to determine VO₂peak and concentric MAP (cMAP), followed by six functional performance assessments.

The training protocol consisted of three consecutive 4-week phases:

1. Familiarization Phase (Weeks 2-5)
2. Initial Training Phase (Weeks 6-9)
3. Progressive Training Phase (Weeks 10-13) with increased training intensity.

At the first and final visits, participants underwent a concentric incremental cycling test to determine VO₂peak and cMAP. The test began with a standardized 2-minute warm-up at 30 watts (W) and a cadence of 60 revolutions per minute (rpm). The workload was then increased every minute by 15 W for women and 20 W for men until volitional exhaustion.

Participants were instructed to maintain a cadence above 60 rpm and were verbally encouraged throughout the test.

The 12-week training intervention was structured into three consecutive phases: (1) familiarization, (2) initial training, and (3) progressive training. All participants completed two supervised sessions per week, either on a recumbent eccentric ergometer (Cyclus 2, RBM Elektronik-Automation GmbH, Germany) or a seated concentric cycle ergometer (Technogym, Italy), depending on group allocation.

1. Phase 1 (T1) - Familiarization (Weeks 2-5) During the familiarization phase, all groups completed work-matched sessions adapted to their respective contraction modality (eccentric or concentric cycling). Based on the findings of Lipski et al., a conversion ratio of 1.5 was used to estimate eccentric MAP (eMAP) from cMAP, such that 100% eMAP was considered equivalent to 150% of cMAP.

   Training intensity and duration were progressively increased across the four weeks. Participants began with 5 minutes of cycling at 30% of their cMAP and progressed to 30 minutes by the end of the phase.
2. Phase 2 (T2) - Initial Training (Weeks 6-9)

   In the second phase, all groups trained at an intensity equivalent to 80% of their modality-specific MAP for 30 minutes per session:
   * EI Group: 10 x 2' training/1' rest at 120% of cMAP (~80% of eMAP)
   * EC Group: 30' at 80% of cMAP
   * CI Group: 10 x 2' training/1' rest at 80% of cMAP
3. Phase 3 (T3) - Progressive Training (Weeks 10-13)

Training intensity was further increased to 90% of each group's modality-specific MAP:

* EI Group: 10 x 2' training/1' rest at 135% of cMAP (~90% of eMAP)
* EC Group: 30' at 90% of cMAP
* CI Group: 10 x 2' training/1' rest at 90% of cMAP This progressive overload aimed to enhance aerobic capacity and muscular adaptations in a contraction-specific manner. All sessions remained isocaloric and time-matched across groups to allow for valid comparisons.

Heart rate, rating of perceived exertion, cognitive demand / fatigue and muscle soreness were monitored during each training session.

A battery of six functional tests was performed pre- and post-intervention to evaluate intra-group improvements and inter-group differences. All tests were administered by the same trained evaluator to minimize inter-rater variability. Standardized instructions and verbal encouragement were provided to ensure consistency across participants. These tests include : maximal isometric force, handgrip strength, balance, ten times sit-to-stand time, timed up and go and six-minute walking test.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary people (less than 3 hours of physical activity a week)
* No smoker

Exclusion Criteria:

* Pain or injury in the 6 previous months in the lower limbes
* Presenting an uncontrolled chronic condition
* Presenting cardiovascular issues

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Maximal Isometric Force | At enrollment and at the end of treatment at 14 weeks
  Maximal isometric knee extensors strength of the dominant leg was assessed using a MicroFET2 handheld dynamometer (Hoggan Scientific, USA) secured to an immovable frame. Participants were seated with hips at 85° and knees at 90° flexion. After a warm-up involving five minutes of low-intensity cycling and three submaximal isometric contractions (50-90% effort), participants completed five maximal voluntary contractions, each lasting five seconds with 30 seconds of rest between efforts. The highest recorded value was retained for analysis and expressed in newton-meters (Nm).
Maximal Aerobic Power | At the begining and the end of study (week 1 and 14)
  At the first and final visits, participants underwent a concentric incremental cycling test to determine their maximal aerobic power (expressed in watt (W)). The test began with a standardized 2-minute warm-up at 30 W and a cadence of 60 revolutions per minute (rpm). The workload was then increased every minute by 15 W for women and 20 W for men until volitional exhaustion. The higher value was recorded as their MAP.
  Participants were instructed to maintain a cadence above 60 rpm and were verbally encouraged throughout the test.
Peak oxygen consumption | At the begining and the end of the study (week 1 and 14)
  At the first and final visits, participants underwent a concentric incremental cycling test to determine VO₂ peak (expressed in mililiters per minute per kilogram (mL/min/kg)). The test began with a standardized 2-minute warm-up at 30 watts (W) and a cadence of 60 revolutions per minute (rpm). The workload was then increased every minute by 15 W for women and 20 W for men until volitional exhaustion. The higher value of VO₂ was recorded as their VO₂ peak.
  Participants were instructed to maintain a cadence above 60 rpm and were verbally encouraged throughout the test.
Weight | At the begining and the end of the study (week 1 and 14)
  Study participants were weighed during their first session of participation. This measurement was taken on a Tanita balance and is expressed in kilograms (kg).
Height | At the begining and the end of the study (week 1 and 14)
  Participants were measured during their first session of participation in the study. This measurement was taken using a wall-mounted height gauge and is expressed in meters (m).
Body mass index | At the begining and the end of the study (week 1 and 14)
  The body mass index (BMI) of the participants was calculated based on their previously measured weight and height. The following formula was used: weight (kg)/height (m)², and BMI is expressed in kg/m^2
Body fat index | At the begining and the end of the study (week 1 and 14)
  The body fat percentage of each participant was measured using Tanita scales and expressed as a percentage (%).

SECONDARY OUTCOMES:
Handgrip strength | At week 1 and week 14
  Handgrip strength of the dominant hand was measured using a handheld isometric dynamometer (Takei Hand Grip Dynamometer, Japan). Participants performed three maximal grip trials, with 30 seconds of rest between each trial. During testing, the arm was kept extended along the body without any auxiliary movements. The best value was retained and expressed in kilograms (kg).
Balance error scoring system | Week 1 and 14
  Static balance was assessed using the BESS protocol, which includes three stance positions (double-leg, single-leg, and tandem) performed on both firm and foam surfaces. Each position was held for 20 seconds with eyes closed and hands on hips. Errors, such as opening eyes, lifting hands or losing balance were counted, with a maximum of 10 errors per trial.
Ten times sit to stand test | Week 1 and 14
  Functional lower limb strength and mobility were assessed via the TTSST. Participants began seated with arms crossed over their chest and were instructed to stand up and sit down 10 times as quickly as possible. The test started with a countdown and was timed using a stopwatch. Participants performed 3 trials and the best values was retained for analysis and expressed in seconds (s).
Timed up and go | Week 1 and 14
  Mobility and dynamic balance were assessed using the TUAG test. Participants rose from a seated position, walked three meters, turned 180°, returned to the chair, and sat down, performing a second 180° turn. The time to complete the sequence was recorded with a stopwatch. Participants performed 3 trials and the best values was retained for analysis and expressed in seconds (s).
Six-minute walking test | Week 1 and 14
  Aerobic endurance was evaluated via the 6MWT. Participants were instructed to walk as far as possible in six minutes along a 30-meter indoor track, turning around two cones at either end. HR and RPE were monitored throughout the test. The total distance covered was expressed in meters (m).

OTHER OUTCOMES:
Rating of perceived exertion | Throughout all the training sessions (week 2 to week 13)
  At the end of each training session, participants reported their rating of perceived exertion (RPE) using the Borg RPE scale, ranging from 6 (no exertion) to 20 (maximal exertion)
Heart Rate | Throughout the training sessions, from week 2 to week 15
  Mean and Maximal heart rate (HR) were recorde throughout each training session using a polar sensor ("polar verity sense"). Heart rate is expressed in beats per minute (bpm).
Cognitive demand | At the end of each training session, from week 2 to week 15
  The cognitive demand / fatigue perceived during the training was recorded at the end of each session, using the modified Borg Category-Ratio 10 (CR-10) scale, ranging from 0 (no effort) to 10 (maximal effort).
Perceived muscle soreness in the lower limbs | At the beginning of each training session, from week 2 to week 15
  Perceived muscle soreness in the lower limbs (DOMS) were monitored at the beginning of each training session, using a visual analog scale (VAS) ranging from 0 mm (no soreness) to 200 mm (unbearable soreness).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie HODY, PhD, Study Director — ULiege - Supervisor; Jean-François Kaux, Prof, Study Director — ULiege - Co-supervisor
Locations (1):
- Liege University, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT07189975/Prot_SAP_000.pdf